CLINICAL TRIAL: NCT01476735
Title: A Prospective, Randomized, Single-blind Study Evaluating Individual Approach on Bowel Preparation Quality for Colonoscopy
Brief Title: Individual Approach for Bowel Preparation Before Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Individual bowel preparation
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2011-11

CONDITIONS: Split-dose Bowel Preparation; Polyethylene Glycol Solution; Risk Factors Inadequate Preparation
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- split-dose polyethylene glycol solution (Active Comparator): first dose (1,5 l) of polyethylene glycol solution taken at 6-7.00 in the evening before colonoscopy, second dose (1,5 l) taken at 5.30-6.00 in the morning of a day of colonoscopy; additional bisacodyl taken at 12.00 at the day before colonoscopy
  Interventions: Other: individual preparation for colonoscopy
- Individual preparation for colonoscopy (Active Comparator)
  Interventions: Other: individual preparation for colonoscopy

INTERVENTIONS:
Other: individual preparation for colonoscopy — The volume of polyethylene glycol solution depends on risk factors presented in each patient. Time of administration of second dose will be confirmed according to the time of colonoscopy. In case of constipation an enema before colonoscopy will be administered. All patients will give educational booklet of preparation before colonoscopy

SUMMARY:
This is a prospective, randomized, single-blind study designed to evaluate the influence of individual approach on bowel preparation quality for colonoscopy. The investigators compare split-dose polyethylene glycol solution (PEG, Fortrans, Beaufour Ipsen) to modified split-dose PEG regarding predictors of inadequate preparation for colonoscopy.

DETAILED DESCRIPTION:
Up to 22% of patients are not good prepared for colonoscopy and it is caused of aborted procedures and increased costs. There are identified predictors of inadequate bowel preparation before colonoscopy, but we still don't know if an individual approach improve the quality of preparation.

ELIGIBILITY:
Inclusion Criteria:

* men and women more than 18 years of age undergoing colonoscopy for routine clinical indications
* provided written informed consent

Exclusion Criteria:

* lack of written informed consent or inability to provide informed consent or refusal to consent to the study
* pregnancy and breast feeding
* known allergy to PEG or bisakodyl
* presence of serious conditions such as severe cadiac, renal or metabolic diseases, major psychiatric illness or end-stage cancer disease requiring taking narcotic drugs
* colonoscopy performed under conscious sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the index of preparation quality for the whole colon | 24 hours
  the percentage of patients with adequate bowel preparation; adequate preparation is defined as excellent, good and fair, inadequate is defined as poor or unprepared colon according to the Ottawa bowel preparation scale

SECONDARY OUTCOMES:
compliance safety | 24 hours
  number of patients with completion of preparation number of patients with side effects of preparation in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Regula, MD, PhD, Study Director — Maria Sklodowska-Curie Memorial cancer Center, Institute of Oncology, Warsaw, Poland; Michal F. Kaminski, MD, Study Chair — Maria Sklodowska-Curie Memorial cancer Center, Institute of Oncology, Warsaw, Poland; Dorota Wretowska, MD, Principal Investigator — Maria Sklodowska-Curie Memorial cancer Center, Institute of Oncology, Warsaw, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial cancer Center, Institute of Oncology, Warsaw, Poland